CLINICAL TRIAL: NCT00010205
Title: Phase I Trial Of Benzoylphenylurea (NSC#639829) In Advanced Malignancy
Brief Title: Benzoylphenylurea in Treating Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02375; UMGCC 0038; U01CA069854 (NIH); CDR0000068455 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

ARMS (1):
- Treatment (benzoylphenylurea) (Experimental): Patients receive oral benzoylphenylurea weekly for 6 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of benzoylphenylurea until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity.
  Interventions: Drug: benzoylphenylurea; Other: pharmacological study

INTERVENTIONS:
Drug: benzoylphenylurea — Given orally
  Other Names: BPU
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of benzoylphenylurea in treating patients with advanced cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the dose-limiting toxicity and the maximum tolerated dose of benzoylphenylurea in patients with advanced malignancy.

II. Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral benzoylphenylurea weekly for 6 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of benzoylphenylurea until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy

  * Metastatic or unresectable
  * No standard curative or palliative measures exist or are ineffective
* Brain metastases allowed provided 1 of the following criteria is met:

  * Lesions were previously treated with surgery, radiotherapy, or chemotherapy AND are currently asymptomatic AND no steroid therapy or antiseizure medication within the past 2 weeks
  * Untreated, asymptomatic metastases AND no requirement for steroid therapy or antiseizure medication
* Performance status - ECOG 0-2
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal
* Albumin at least 3.0 mg/dL
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* No prior allergic reactions to compounds of similar chemical or biologic composition to benzoylphenylurea
* No neuropathy greater than grade 1
* No other uncontrolled medical or psychiatric illness that would preclude study compliance
* No ongoing or active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Prior immunotherapy allowed
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* At least 2 weeks since steroids for CNS disease
* At least 4 weeks since prior radiotherapy and recovered
* Prior surgery allowed
* At least 2 weeks since antiseizure medications for CNS disease
* More than 7 days since prior CYP3A4 or CYP2D6 inhibitors
* More than 7 days since prior CYP3A4 inducers
* No concurrent CYP3A4 or CYP2D6 inhibitors
* No concurrent CYP3A4 inducers
* No other concurrent investigational agents
* No concurrent combination anti-retroviral therapy for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-12; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) defined as the highest dose level where 0/6 or 1/6 patients experience dose-limiting toxicity (DLT) as assessed by CTCAE version 3.0 | 8 weeks
DLT defined as grade 3 or worse non-hematologic and sustained (> 5 days) grade 3 hematologic toxicity or grade 4 hematologic toxicity of any duration, and the moderate toxicity is grade 2 toxicity as assessed by CTCAE version 3.0 | 8 weeks
Pharmacokinetics of benzoylphenylurea | At baseline, at 0.5, 1.0, 1.5, 2, 4, 6, 8, 24, 48, 72, and 96 hours (weeks 1 and 6)
  Relationships between drug exposure and toxicity, efficacy, and biological endpoints will be explored using univariate and multivariate analysis techniques.

SECONDARY OUTCOMES:
Response (complete and partial response) rate | Up to 7 years
  Response rate will be evaluated for all patients with measurable disease and will be obtained by dividing the total number of responses by all patients with measurable disease and reported with 95% confidence intervals.
Survival | From the date of first treatment until death or last follow-up, assessed up to 7 years
  The median and landmark survivals will be estimated utilizing the Kaplan- Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Edelman, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States